CLINICAL TRIAL: NCT01208714
Title: Endovascular Treatment Versus Optimal Medical Treatment of Atherosclerotic Renal Artery for Preserving Renal Function of the Ischemic Kidney.
Brief Title: Medical and Endovascular Treatment of Atherosclerotic Renal Artery Stenosis (METRAS Study)
Acronym: METRAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Padova (Other)
Responsible Party: Gian Paolo Rossi, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GPR-METRAS
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-09

CONDITIONS: Renal Artery Stenosis
Keywords: Renal artery stenosis; Atherosclerosis; Arterial hypertension; Percutaneous renal angioplasty; Stenting
MeSH Terms: conditions — Renal Artery Obstruction; Atherosclerosis; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- revascularization (Active Comparator): The patients randomized to this treatment will undergo PTA with stenting of the renal artery.
  Interventions: Procedure: revascularization
- medical therapy (Active Comparator): The patients randomized to this treatment will undergo optimal medical therapy
  Interventions: Drug: Optimal medical therapy

INTERVENTIONS:
Drug: Optimal medical therapy — Optimal medical therapy, including optimal antihypertensive therapy as defined by ESH/ESC Guidelines Mancia G. J Hypertens 2007; 25: 1105), antiplatelet and, if necessary, hypolipemic and hypoglycemic treatment.
  All patients will receive antiplatelet treatment with the same dose of aspirin (100 mg o.d.) or ticlopidine (250 mg b.i.d) if intolerant ASA, or clopidogrel (75 mg o.d.), if intolerant to ASA and ticlopidine, throughout the study period. LDL-cholesterol will be lowered to below 100 mg/dl, homocysteine if elevated will be lowered and treatment for diabetes will be optimized (HbA1c < 6.5%).
  Arms: medical therapy
Procedure: revascularization — The patients randomized to this treatment will undergo digital scan angiography (DSA) and PTA with stenting of the renal artery. PTA will be performed at the ostium or at truncular level. Stenoses involving more distal arterial vessels will be recorded and considered for data analysis but will not be treated. The patients randomized to revascularization will continue on their antihypertensive drug regimen. The dose and number of drugs will be down-titrated with the aim of pursuing the target BP values.
  Other Names: Device: Palmaz Genesis stent on Cordis AMIIA delivery system
  Arms: revascularization

SUMMARY:
Renal atherosclerotic stenosis (RAS) is a prevalent cause of secondary hypertension (HT). Since there are still uncertainties as to whether and in what patients revascularization by means of percutaneous renal angioplasty (PTRAS) should be pursued, we designed a study exploiting an optimized patient selection strategy and using hard experimental endpoints to unravel these uncertainties.

Primary objective: to determine if revascularization by means of PTRAS is superior or equivalent to optimal medical treatment for preserving glomerular filtration rate in the ischemic kidney as assessed by 99mTcDTPA sequential renal scintiscan.

Secondary objectives: to determine if the two treatments are equivalent in lowering blood pressure (BP), preserving overall renal function and regressing damage in the target organs of hypertension.

Design: prospective multicenter randomized, unblinded two-arm study.

Eligible patients will have clinical and/or radiological evidence of unilateral or bilateral RAS, defined by stenosis of the proximal portion of the renal artery and its main bifurcations at angioCT. Duplex scan will exclude nephroangiosclerosis as the latter could bias the assessment of the outcome of revascularization.

Inclusion criteria. RAS affecting the main renal artery or its major branches at angio-CT either > 70% or, if < 70 with post-stenotic dilatation.

Renal function will be assessed with 99mTc-DTPA renal scintigraphy.

Sample size (30 patients per arm) was calculated to have a 90% power to detect a difference in means of GFR in the vascularized (or control untreated kidney) of 7.5 ml/min.

Arms

1. Revascularization: digital scan angiography and PTA with stenting of the renal artery at the ostium or at truncular level, plus optimal medical therapy.
2. Medical therapy: the drug regimen that had been optimized during the run-in period.

Experimental endpoints:

The absolute value of GFR assessed by 99TcDTPA in the ischemic kidney will be used as quantitative variable and compared between groups at each time point. A categorical definition of kidney loss, defined as a GFR in the ischemic kidney of < 5 ml/min, will be also used and the rate of achievement of such endpoint will be compared.

Duration: 5 years.

DETAILED DESCRIPTION:
Background Renal atherosclerotic stenosis (RAS) is an increasingly prevalent causes of secondary hypertension (HT), and is becoming one of the first causes of end-stage renal failure requiring renal replacement therapy in an aging population. Atherosclerotic RAS is associated with a high cardiovascular risk profile leading to a considerable excess rate of morbidity and mortality from stroke, coronary heart and peripheral vascular disease.

Recent advances in antihypertensive drug therapy and in intensive risk factor management prompted the undertaking of prospective randomized trials that compared percutaneous renal angioplasty (PTRAS) with medical therapy. Unexpectedly, these trials failed to show compelling benefits of revascularization when added to effective medical therapy. However, they had serious limitations, which raised a number of criticisms, and limited to weight of their conclusions. Hence, clinicians are still left with uncertainties as to whether and in what patients revascularization should be pursued.

It is conceivable that only a study design exploiting an optimized patient selection strategy and a use of hard experimental endpoints could resolve these uncertainties and thus lead to a better clinical management of the increasing population with atherosclerotic RAS.

Objectives. The primary objective of the METRAS study is to determine if revascularization by means of PTRAS is superior or equivalent to optimal medical treatment for preserving glomerular filtration rate in the ischemic kidney as assessed by 99TcDTPA sequential renal scintiscan.

Secondary objectives (see appropriate section) will be to determine if the two treatments are equivalent in lowering blood pressure (BP), preserving overall renal function and regressing damage in the target organs of hypertension.

Design: prospective multicenter randomized, unblinded two-arm study. Enrolment. Eligible patients entail adult hypertensive of both genders with clinical and/or radiological evidence of unilateral or bilateral RAS. Clinical evidence of RAS will be unexplained renal dysfunction (GFR < 60 ml/min), uncontrolled or refractory hypertension (defined as resistant to lifestyle measures and to at least 3 drugs including a diuretic in adequate doses with failure in lowering systolic and diastolic BP to goal) and/or significant worsening of renal function (20% increase of serum creatinine) after administration of ACE inhibitors and/or an abdominal bruit and/or evidence of atherosclerotic involvement of other sites.

Radiological evidence of atherosclerotic RAS will be defined by stenosis of the proximal portion of the renal artery and its main bifurcations at angioCT. Besides Angio-CT, patients will undergo Duplex scan to exclude nephroangiosclerosis as the latter could bias the assessment of the outcome of revascularization.

Eligible subjects will be offered participation to the METRAS study and have to sign an informed written consent.

Inclusion criteria: angio-CT evidence of RAS affecting the main renal artery or its major branches > 70% or, if < 70 with post-stenotic dilatation Exclusion criteria: see dedicated section.

Run-in. Eligible patients will undergo a 4-week run-in period during which BP treatment, LDL-cholesterol, homocysteine and glycemic control will be optimized.

All patients will receive antiplatelet treatment with aspirin or ticlopidine if intolerant ASA, or clopidogrel, if intolerant to ASA and ticlopidine, throughout the study period.

AngioCT will be performed to assess the abdominal aorta and renal artery anatomy and pathology. RAS localization will be assessed blindly by 2 experienced radiologists. Precautions will be adopted to minimize the chances of worsening renal function with angioCT.

99mTc-DTPA renal scintigraphy will be performed on 2 consecutive days, before and after captopril administration, according to available guidelines.

Treatment with ACEI/ARB will be stopped for 3-7 days (depending on drug half-life) before the scintigraphy. If ACEI withdrawal will be held to be unsafe, the captopril scintigraphy will be omitted and only baseline 99mTc-DTPA scintigraphy will be performed.

All on-site measurements from imaging will be validated by a core laboratory at the University of Padova.

Renal function will be assessed with MDRD formula and the reciprocal of creatinine.

Target organ damage (TOD). Transthoracic echocardiogram with Doppler with assessment of LV mass index, relative thickness, the E/A wave peak flow velocity rate and tissue Doppler will be used to detect changes in LV remodeling and diastolic filling. Measurement of pulse wave velocity, and augmentation index will be used to follow the changes in aortic stiffness and vascular damage.

BP. Clinic and ambulatory BP monitoring (ABPM) will be performed to evaluate the BP changes in each treatment arm. ABPM will be used to determine the BP variability (smoothness index) during day and night.

Randomization. A matching algorithm considering both the RI and the presence of unilateral/bilateral stenosis will be used to randomly assign patients to the 2 treatment arms. This randomization strategy will allow us to obtain patients with similar distribution of RI and an equal number of the patients with unilateral and bilateral stenosis in each treatment arm.

Sample size. Power calculation (nQuery Vers, 6.0, Statistical Solutions) showed that assuming a 16% drop-out rate, a common standard deviation of 8.0 ml/min, an equal sample size in each treatment arm, using a two group t-test with a 0.05 2-sided significance level, with 30 patients per arm our study will have a 90% power to detect a difference in means of GFR in the vascularized (or control untreated kidney) of 7.5 ml/min.

Treatment arms

1. Revascularization. The patients randomized to this treatment will undergo digital scan angiography (DSA) and PTA with stenting of the renal artery. PTA will be performed at the ostium or at truncular level. Stenoses involving more distal arterial vessels will be recorded and considered for data analysis but will not be treated. The patients randomized to revascularization will continue on their antihypertensive drug regimen. The dose and number of drugs will be down-titrated with the aim of pursuing the target BP values.
2. Medical therapy The patients randomized to medical treatment will continue only on the antihypertensive drug regimen that had been optimized to reach the BP goal during the run-in period.

Experimental endpoints. The absolute value of GFR assessed by 99TcDTPA in the ischemic kidney will be used as quantitative variable and compared between groups at each time point. Moreover, for the purpose of the Cox regression analysis a categorical definition of kidney loss, defined as a GFR in the ischemic kidney of < 5 ml/min, will be used and the rate of achievement of such endpoint will be compared.

Potential confounders. To minimize the untoward effect of differences in CV risk anti-platelet, lipid-lowering, and antidiabetic agents, when needed, will be given to all patients, and maintained at the same dosage achieved at the end of the run-in period throughout the study. The possible unbalanced distribution of confounders between treatment arms will be handled by calculating the propensity score (8, 9) and entering it in the Cox regression analysis.

Follow-up. Visits will be scheduled at 1, 3, 6, 12 and 24 months after revascularization or beginning of the medical therapy. The study will then continue in an observational setting with outpatient visits scheduled at 6-month intervals for 5 years.

Data collection. Data will be collected using specifically designed database and forms (created in Open Clinica; http://www.openclinica.org); they will be monitored in real time and then analyzed at the core laboratory.

Statistical analysis. Comparison of GFR in the ischemic kidney between groups (revascularization vs. medical therapy) at each time point will be performed using t-test, repeated measure ANOVA with adjustment of potential confounders, Cox regression model for loss of kidney function as defined above. Sub-group analysis (comparison unilateral vs bilateral stenosis) will be similarly undertaken. ROC curves will be used to determine if the baseline 99mTc DTPA scintiscan-derived indexes can predict the outcome of treatment using the changes in GFR over time as reference. Bland-Altman plot and analysis will be used to compare the estimate of GFR obtained using cystatin using the overall (right and left kidneys) GFR as reference.

Multivariate techniques and on the propensity score, which considers all relevant covariables that will differ between the revascularization and the medical treatment rate group, will be used to avoid the untoward effect of a possible unbalanced distribution of confounders between treatment arms (D'Agostino RB, Jr. Circulation 2007; Maiolino G. JCEM 2008).

Expected results. The Metras study will clarify whether renal revascularization by means of PTRAS associated with optimal medical therapy is superior or equivalent to optimal medical treatment alone in preventing deterioration of renal function, as assessed as GFR in the ischemic kidney.

A previous study by Radermacher et al suggested that the presence of irreversible renal microvascular changes, e.g. nephroangiosclerosis, could prevent the patients from having benefit with revascularization. In fact an intrarenal resistance index (RI) > 0.80 at the Doppler analysis was claimed to predict no improvement of BP or renal function, as assessed by measuring the creatinine clearance. However, the latter is an index of global function, and therefore provides no information on the GFR of the ischemic kidney.

This study, by randomizing patients for matching RI values, is expected to clarify whether endovascular treatment can slower GFR loss even in the patients with nephroangiosclerosis.

Moreover, by meeting its secondary endpoints it will help clarifying some clinically relevant issues as the BP lowering, the rate of renal and major cardiovascular events, and the change in quality of life with/without endovascular treatment in patients with atherosclerotic RAS.

Duration of the study. The METRAS Study will last for 5 years. This time interval is expected to be sufficient to register renal and major cardiovascular events.

Centers. This study will be performed within the Italian Society of Arterial Hypertension (SIIA) to achieve randomization of the number of patients needed to provide significant power to the study.

A core laboratory in Padova will adjudicate the eligible patients and will randomize patients.

Conclusions and Perspectives. The METRAS Study has been designed to provide a conclusive answer to a very debated question: is angioplasty combined with stenting and associated with optimal medical therapy equivalent to the optimal medical treatment alone in preventing deterioration of renal function, assessed as GFR in the ischemic kidney? A novel approach, consisting in evaluating deterioration of renal function, as assessed as GFR in the ischemic kidney, rather than the overall GFR, will clarify if PTRAS can protect a kidney with stenotic artery from functional declining.

ELIGIBILITY:
Inclusion Criteria:

* RAS affecting the main renal artery or its major branches at angio-CT either > 70% or, if < 70 with post-stenotic dilatation AND
* resistance index (RI) < 0.55 or > 0.55 but < 0.80 with evidence of intrarenal heterogeneity of the RI as revealed by a CV > 10% in the RI across the upper, mid and lower third of each kidney.

Exclusion Criteria:

* refusal to participate to study,
* previous endovascular or surgical treatment of RAS,
* fibromuscular RAS,
* planned or actual pregnancy, or childbearing potential without measures adequate to prevent pregnancy,
* life expectancy < 2 years,
* patient currently participating in another trial possibly influencing the safety of the patient and/or the outcomes of the study,
* co-morbid conditions limiting participation and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Glomerular filtration rate in the ischemic kidney after revascularization by means of percutaneous renal angioplasty (PTRAS) or optimal medical treatment. | 24 months
  The Primary Objective of the study is to determine if revascularization by means of PTRAS is superior or equivalent to optimal medical treatment for preserving glomerular filtration rate in the ischemic kidney as assessed by 99TcDTPA sequential renal scintiscan

SECONDARY OUTCOMES:
Lowering blood pressure after revascularization by means of percutaneous renal angioplasty (PTRAS) or optimal medical treatment. | 1, 3, 6, 12, 24, 36, 48 and 60 months
  One secondary objective of the study is to determine if the two treatments (revascularization by means of percutaneous renal angioplasty (PTRAS) or optimal medical treatment) are equivalent in lowering blood pressure after revascularization by means of percutaneous renal angioplasty (PTRAS) or optimal medical treatment.
Preserving overall renal function after revascularization by means of percutaneous renal angioplasty (PTRAS) or optimal medical treatment. | 1, 3, 6, 12, 24, 36, 48 and 60 months
  One secondary objective of the study is to determine if the two treatments (revascularization by means of percutaneous renal angioplasty (PTRAS) or optimal medical treatment) are equivalent in preserving overall renal function, as assessed by total estimated GFR, the reciprocal of serum creatinine, and indexes of Ca2+ and PO43- metabolism.
Regression of damage in the target organs of hypertension, including cardiac hypertrophy, microalbuminuria and aortic stiffness after revascularization by means of percutaneous renal angioplasty (PTRAS) or optimal medical treatment. | 1, 3, 6, 12, 24, 36, 48 and 60 months
  One secondary objective of the study is to determine if the two treatments (revascularization by means of percutaneous renal angioplasty (PTRAS) or optimal medical treatment) are equivalent in tregressing damage of the target organs of hypertension, including cardiac hypertrophy, microalbuminuria and aortic stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Paolo Rossi, MD, FACC, Study Director — Dept Clinical and Experimental Medicine (DMCS), University Hospital of Padova, Italy
Locations (1):
- Dept. Clinical and Experimental Medicine, University of Padova, Italy, Padua, Italy

REFERENCES:
- [Background] Cheung CM, Hegarty J, Kalra PA. Dilemmas in the management of renal artery stenosis. Br Med Bull. 2005 Sep 7;73-74:35-55. doi: 10.1093/bmb/ldh049. Print 2005. PMID 16148190
- [Background] Guo H, Kalra PA, Gilbertson DT, Liu J, Chen SC, Collins AJ, Foley RN. Atherosclerotic renovascular disease in older US patients starting dialysis, 1996 to 2001. Circulation. 2007 Jan 2;115(1):50-8. doi: 10.1161/CIRCULATIONAHA.106.637751. Epub 2006 Dec 18. PMID 17179020
- [Background] Plouin PF, Chatellier G, Darne B, Raynaud A. Blood pressure outcome of angioplasty in atherosclerotic renal artery stenosis: a randomized trial. Essai Multicentrique Medicaments vs Angioplastie (EMMA) Study Group. Hypertension. 1998 Mar;31(3):823-9. doi: 10.1161/01.hyp.31.3.823. PMID 9495267
- [Background] Bax L, Mali WP, Buskens E, Koomans HA, Beutler JJ, Braam B, Beek FJ, Rabelink TJ, Postma CT, Huysmans FT, Deinum J, Thien T, Schultze Kool LJ, Woittiez AJ, Kouwenberg JJ, van den Meiracker AH, Pattynama PM, van de Ven PJ, Vroegindeweij D, Doorenbos CJ, Aarts JC, Kroon AA, de Leeuw PW, de Haan MW, van Engelshoven JM, Rutten MJ, van Montfrans GA, Reekers JA, Plouin PF, La Batide Alanore A, Azizi M, Raynaud A, Harden PN, Cowling M; STAR Study Group. The benefit of STent placement and blood pressure and lipid-lowering for the prevention of progression of renal dysfunction caused by Atherosclerotic ostial stenosis of the Renal artery. The STAR-study: rationale and study design. J Nephrol. 2003 Nov-Dec;16(6):807-12. PMID 14736007
- [Background] ASTRAL Investigators; Wheatley K, Ives N, Gray R, Kalra PA, Moss JG, Baigent C, Carr S, Chalmers N, Eadington D, Hamilton G, Lipkin G, Nicholson A, Scoble J. Revascularization versus medical therapy for renal-artery stenosis. N Engl J Med. 2009 Nov 12;361(20):1953-62. doi: 10.1056/NEJMoa0905368. PMID 19907042
- [Background] White CJ. Kiss my astral: one seriously flawed study of renal stenting after another. Catheter Cardiovasc Interv. 2010 Feb 1;75(2):305-7. doi: 10.1002/ccd.22416. No abstract available. PMID 20095015
- [Background] van Jaarsveld BC, Pieterman H, van Dijk LC, van Seijen AJ, Krijnen P, Derkx FH, Man in't Veld AJ, Schalekamp MA. Inter-observer variability in the angiographic assessment of renal artery stenosis. DRASTIC study group. Dutch Renal Artery Stenosis Intervention Cooperative. J Hypertens. 1999 Dec;17(12 Pt 1):1731-6. doi: 10.1097/00004872-199917120-00010. PMID 10658939
- [Background] Maiolino G, Cesari M, Sticchi D, Zanchetta M, Pedon L, Antezza K, Pessina AC, Rossi GP. Plasma adiponectin for prediction of cardiovascular events and mortality in high-risk patients. J Clin Endocrinol Metab. 2008 Sep;93(9):3333-40. doi: 10.1210/jc.2007-2405. Epub 2008 Aug 12. PMID 18697874
- [Background] D'Agostino RB Jr. Propensity scores in cardiovascular research. Circulation. 2007 May 1;115(17):2340-3. doi: 10.1161/CIRCULATIONAHA.105.594952. No abstract available. PMID 17470708
- [Background] Radermacher J, Chavan A, Bleck J, Vitzthum A, Stoess B, Gebel MJ, Galanski M, Koch KM, Haller H. Use of Doppler ultrasonography to predict the outcome of therapy for renal-artery stenosis. N Engl J Med. 2001 Feb 8;344(6):410-7. doi: 10.1056/NEJM200102083440603. PMID 11172177